CLINICAL TRIAL: NCT07201233
Title: Clinical Study on the Safety and Efficacy of Unrelated Umbilical Cord Blood Infusion in Treating Bone Marrow Suppression After Chemotherapy in Elderly Patients With Myelodysplastic Syndrome (MDS) and Acute Myeloid Leukemia (AML) .
Brief Title: Clinical Study on the Safety and Efficacy of Umbilical Cord Blood Infusion in Treating Bone Marrow Suppression .
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong Qilu Stem Cells Engineering Co., Ltd. (Industry)
Collaborators: Tianjin Medical University General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCB-2025
Record Dates: First submitted 2025-09-19; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Bone Marrow Suppression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Umbilical cord blood (Experimental)
  Interventions: Biological: Umbilical cord blood

INTERVENTIONS:
Biological: Umbilical cord blood — Umbilical cord blood transfusion should be performed 24 hours to 2 weeks after chemotherapy. One to multiple units of cord blood can be applied, and the minimum interval between two cord blood transfusions should be 2 weeks.

SUMMARY:
The clinical study aims to evaluate the safety and efficacy of umbilical cord blood transfusion in treating bone marrow suppression after chemotherapy in elderly patients with MDS and AML

DETAILED DESCRIPTION:
The clinical study aims to evaluate the safety and efficacy of umbilical cord blood （HLA typing 0-3/10 match, TNC ≥ 3×10^7/kg）transfusion in treating bone marrow suppression after chemotherapy in elderly patients with MDS and AML，UCB can be applied in one to multiple doses, and the minimum interval between two cord blood transfusions should be 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 1) Ages 60-80 years , gender unlimited;
* 2) Patients clinically diagnosed with MDS or AML;
* 3) Completed chemotherapy and clinically diagnosed with bone marrow suppression grade 2 or above;
* 4) Patients with no severe impairment of liver and kidney function (total bilirubin (TBIL): ≤ 1.5×ULN; ALT or AST: ≤ 2.5×ULN; Alkaline phosphatase: ≤ 3×ULN; Serum creatinine: ≤ 1.5×ULN);
* 5) Normal cardiac function;
* 6) Patients with ECOG 0-2;
* 7) Patients or their families have been informed and voluntarily signed a written informed consent form.

Exclusion Criteria:

* 1) Other factors that may cause abnormalities in white blood cells and neutrophils, such as concurrent infections, invasive procedures, etc.
* 2)Presence of interstitial lung disease, non-infectious pneumonia, or uncontrolled systemic diseases (such as diabetes, hypertension, pulmonary fibrosis, and acute pneumonia, etc.). Any unstable systemic diseases: including but not limited to unstable angina, cerebrovascular accident or transient ischemic attack (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), congestive heart failure (New York Heart Association NYHA classification ≥ III,), severe arrhythmias requiring medication, liver, kidney, or metabolic diseases.
* 3) Any other uncontrolled active diseases that may interfere with participation in the trial;
* 4) Concurrent diagnosis of malignant tumors in other organs;
* 5) Concurrent diagnosis of other hematological disorders;
* 6) Inability to understand or comply with the study protocol;
* 7) Individuals deemed unsuitable for participation in this trial by the investigator.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with bone marrow suppression grade < II. | Tests should be conducted every two days after umbilical cord blood transfusion, for a maximum of 30 days.
  Calculate the percentage of patients with bone marrow suppression grade < II based on recorded hematological parameters.
hematological parameters like hemoglobin level(Hb) | Tests should be conducted every two days after umbilical cord blood transfusion, for a maximum of 30 days.
  Monitor and record hemoglobin level(g/L), every 2 days in patients, and maintain a record.
hematological parameters like white blood cell count(WBC) | Tests should be conducted every two days after umbilical cord blood transfusion, for a maximum of 30 days.
  Monitor and record white blood cell count( 10⁹/L)every 2 days in patients, and maintain a record.
hematological parameters like platelet count(PLT) | Tests should be conducted every two days after umbilical cord blood transfusion, for a maximum of 30 days.
  Monitor and record platelet count ( 10⁹/L)every 2 days in patients, and maintain a record.
hematological parameters like neutrophil count(ANC) | Tests should be conducted every two days after umbilical cord blood transfusion, for a maximum of 30 days.
  Monitor and record neutrophil count ( 10⁹/L)every 2 days in patients, and maintain a record.

SECONDARY OUTCOMES:
Incidence of bleeding | Up to 30 days after umbilical cord blood treatment
  To investigate the efficacy characteristics, percentages will be calculated.
Incidence of infection | Up to 30 days after umbilical cord blood treatment.
  To investigate the efficacy characteristics, percentages will be calculated.

IPD SHARING:
Plan to Share IPD: No